CLINICAL TRIAL: NCT03967015
Title: Developing Low-Cost Universal Malnutrition Screening for Low Income Countries - the MAMMS Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Christine McGrath, Assistant Professor, School of Public Health, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00006221
Record Dates: First submitted 2019-05-13; First posted 2019-05-29 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Child Malnutrition
Keywords: Mobile Health; Kenya; Randomized Controlled Trial
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Administered Malnutrition Monitoring System (MAMMS) (Experimental): Participants randomized to the MAMMS arm will receive MUAC training and nutritional education at enrollment. A short message service (SMS) message will be sent at 7 days following enrollment asking them to measure and send their child's MUAC. Weekly SMS messages asking for the child's MUAC measurement will be sent every 7 days until the last study visit at 180 days following enrollment.
  Interventions: Other: Maternal Administered Malnutrition Monitoring System (MAMMS)
- Standard of care (SOC) (No Intervention): Participants randomized to the standard of care (SOC) arm will receive the same MUAC training and nutritional education as mothers in the MAMMS arm. To accurately simulate community malnutrition outreach programs, no SMS message will be sent to participants in this arm.

INTERVENTIONS:
Other: Maternal Administered Malnutrition Monitoring System (MAMMS) — Participants randomized to the MAMMS arm will be provided with two insertion MUAC tapes that are UNICEF color coded and numbered to 1 mm gradations to take home with them. Participants will receive a weekly SMS asking them to measure and send their child's MUAC via SMS. SMS messages will provide actionable reminders to measure and send the child's MUAC. Both the SMS sent to the participant and SMS responses sent by the participant to the MAMMS system will be free of charge. Study staff will screen all SMS measurements returned to the MUAC system for identification of malnutrition.
  Arms: Maternal Administered Malnutrition Monitoring System (MAMMS)

SUMMARY:
Acute malnutrition affects 52 million children, costs $2.1 trillion globally, and contributes to 45% of deaths among children under five years of age. Affordable home-based treatments can prevent many of these deaths, with success rates over 97.5% if malnutrition is identified early. If identified late, treatment failure rates increase to 16%. Malnutrition programs currently rely on community health volunteers to screen children, which can lead to high costs, low screening coverage, and late identification. Mid upper arm circumference (MUAC) is the preferred community malnutrition screening tool. Training mothers to use MUAC tapes to monitor their child's nutritional status through a short message service (SMS) mobile health system could increase screening coverage and facilitate rapid engagement with nutritional services where necessary. The investigators propose to test the "Maternal Administered Malnutrition Monitoring System" (MAMMS) in a randomized controlled trial in Kenya. Participants will be taught to measure their child's MUAC at 6 or 9-month immunization visits and during 6-month follow up the participants will receive a weekly SMS prompting them to measure and send their child's MUAC to a computer system which will alert a health worker when a child with malnutrition is identified. This scalable system could enable nutrition programs to optimize screening coverage, leading to early identification of malnutrition, lower costs and a reduction in under-five mortality.

DETAILED DESCRIPTION:
Acute malnutrition is a critical driver of pediatric mortality that must be addressed to achieve global child health targets. Provision of ready-to-use therapeutic foods (RUTF) and nutritional counselling in the community is a highly effective method of preventing deaths among malnourished children. However, UNICEF estimates that only 17% of malnourished children receive treatment. Among children who are treated, the diagnosis of acute malnutrition is often made late in their disease when the risk of complications and death increases from 2.5% to 16%. Increasing the coverage and frequency of nutritional screening to identify malnourished children earlier in the disease process is a critical step toward achieving global child health goals.

Mid-upper arm circumference (MUAC) is the preferred community malnutrition screening tool. Recent evidence comparing MUAC measurements taken by mothers and community health workers showed that mothers can accurately measure their child's MUAC and identify malnutrition. Yet, there is no pragmatic method of linking these mothers to the nutritional care that malnourished children require. Training and supporting mothers to use MUAC tapes to monitor their child's nutritional status through a two-way short message service (SMS) mobile health system could dramatically increase the coverage of malnutrition screening and facilitate rapid engagement with nutritional service where necessary.

This randomized controlled trial will test the "Maternal Administered Malnutrition Monitoring System" (MAMMS) in western Kenya. Participants will be taught to measure their child's MUAC at 6 or 9-month immunization visits and during 6-month follow up participants will receive weekly SMS messages prompting them to measure and send their child's MUAC to a computer system which will alert a health worker when a child with malnutrition is identified. This scalable childhood growth monitoring system could enable nutrition programs in low and middle income countries to optimize screening coverage, leading to early identification of malnutrition, lower costs and a reduction in global under-five mortality. The study aims to:

Aim 1: Determine if MAMMS leads to earlier identification and recovery from acute malnutrition (MUAC <12.5cm).

Hypothesis 1.1: Children randomized to MAMMS who develop acute malnutrition will be identified earlier than children in the control arm.

Hypothesis 1.2: Children randomized to MAMMS who develop acute malnutrition will be more likely to successfully complete nutritional rehabilitation (defined as no death, no hospitalization, no severe acute malnutrition, and resolution of moderate malnutrition within 4 months of diagnosis) than children in the control arm diagnosed with acute malnutrition.

Aim 2: Demonstrate the accuracy of maternal administered MUAC assessments compared to trained community health worker, and the ability of repeated maternal administered MUAC measurements to monitor early childhood growth.

Hypothesis 2.1: Maternally measured MUAC will be strongly correlated with health worker measured MUAC at baseline and during follow-up.

Hypothesis 2.2: A highly sensitive and specific growth trajectory that predicts moderate acute malnutrition can be identified using maternally measured MUAC.

Aim 3: Evaluate the acceptability, feasibility, fidelity and cost per-child-treated of MAMMS relative to standard-of-care nutrition programs.

Hypothesis 3.1: MAMMS will be acceptable and feasible to mothers and health workers.

Hypothesis 3.2: MAMMS will have a substantially lower cost-per-malnutrition case identified than standard screening approaches.

ELIGIBILITY:
Inclusion Criteria:

* Infant is 6-12 months of age and MUAC of 12.5-14.0 cm
* Access to a mobile phone and can provide a mobile phone number
* Planning to remain in the catchment area more than 6 months and willing to return for 6-month follow up visit
* Mother is willing to be randomized to weekly SMS and measure and send weekly infant MUAC via SMS
* Able to read or write or has someone to help them read or write

Exclusion Criteria:

* Infant is currently on treatment for malnutrition
* Inability to provide a mobile phone number
* Mothers that could not read or write and did not have someone to help them read or write

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-08-02 (Estimated); Study Completion 2022-02-03 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of acute malnutrition [mid-upper arm circumference (MUAC) <12.5cm] following randomization | 6 months

SECONDARY OUTCOMES:
Number of children who recover from acute malnutrition (no death, no hospitalization, weight-for-length z-score>-2 and/or MUAC≥12.5cm) among those identified with acute malnutrition (MUAC<12.5cm) following randomization | 4 months
Mean difference in participant and field worker MUAC measures between baseline and outcome assessment | 6 months
Mean change in MUAC between baseline and outcome assessment | 6 months
Proportion of participants in the MAMMS arm that report continued interest in participation in the MAMMS intervention at outcome assessment | 6 months
Proportion of delivered short message service (SMS) messages that the participant responds to | 6 months
Proportion of delivered short message service (SMS) messages that the participant responds to by mobile phone ownership | 6 months
Proportion of delivered short message service (SMS) messages that the participant responds to by participant literacy | 6 months
Mean change in the number of delivered short message service (SMS) messages that the participant responds between baseline and outcome assessment | 6 months
Mean change in the number of delivered short message service (SMS) messages that the participant responds between baseline and outcome assessment by mobile phone ownership | 6 months
Mean change in the number of delivered short message service (SMS) messages that the participant responds between baseline and outcome assessment by participant literacy | 6 months
Mean unit cost per child identified with acute malnutrition (MUAC<12.5cm) following randomization | 6 months
Mean incremental total costs (economic and financial costs) per child identified with acute malnutrition (MUAC<12.5cm) following randomization | 6 months
Mean unit cost per child treated for acute malnutrition among those identified with acute malnutrition (MUAC<12.5cm) following randomization | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine J McGrath, PhD, MPH, Principal Investigator — University of Washington
Locations (3):
- Kenya (3):
  - Homa Bay County Referral Hospital, Homa Bay
  - Nyatike (Macalder) Sub-County Hospital, Macalder
  - Migori County Referral Hospital, Migori

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: IPD that underlie results in a publication will be made publicly available within 6 months of the publication.
Access Criteria: IPD that underlie results in a publication will be made publicly available in an open access repository within 6 months of the publication.

REFERENCES:
- [Derived] Tickell KD, Achieng C, Masheti M, Anyango M, Ndirangu A, Diakhate MM, Yoshioka E, Levin C, Rubin Means A, Choo EM, Ronen K, Unger JA, Richardson BA, Singa BO, McGrath CJ. Family MUAC supported by a two-way SMS platform for identifying children with wasting: the Mama Aweza randomised controlled trial. EClinicalMedicine. 2023 Sep 21;64:102218. doi: 10.1016/j.eclinm.2023.102218. eCollection 2023 Oct. PMID 37781159
- [Derived] Tickell KD, Diakhate MM, Goodman JL, Unger JA, Richardson BA, Rubin Means A, Ronen K, Levin C, Choo EM, Achieng C, Masheti M, Singa BO, McGrath CJ. Impact of a two-way short message service (SMS) to support maternally administered childhood mid-upper arm circumference monitoring and expand malnutrition screening in Kenya: the Mama Aweza trial protocol. BMJ Open. 2020 Sep 22;10(9):e036660. doi: 10.1136/bmjopen-2019-036660. PMID 32963066